CLINICAL TRIAL: NCT00003967
Title: A Phase I Study of Sequential Prolonged Oral Topotecan (IND# 58,131) and Prolonged Oral Etoposide as Second Line Therapy in Ovarian, Peritoneal or Tubal Carcinoma
Brief Title: Topotecan Plus Etoposide in Treating Patients With Recurrent Ovarian, Peritoneal, or Fallopian Tube Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: GOG Foundation (Network)
Purpose: Treatment
Other Study IDs: CDR0000067168; GOG-9807
Record Dates: First submitted 1999-11-01; First posted 2004-03-31 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2008-03

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: recurrent ovarian epithelial cancer; ovarian undifferentiated adenocarcinoma; ovarian mixed epithelial carcinoma; ovarian serous cystadenocarcinoma; ovarian mucinous cystadenocarcinoma; ovarian endometrioid adenocarcinoma; ovarian clear cell cystadenocarcinoma; fallopian tube cancer; primary peritoneal cavity cancer; Brenner tumor
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial; Brenner Tumor | interventions — Etoposide; Topotecan

INTERVENTIONS:
Drug: etoposide
Drug: topotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of topotecan plus etoposide in treating patients who have recurrent ovarian cancer, peritoneal cancer, or fallopian tube cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of sequential prolonged topotecan and prolonged etoposide as second line therapy in patients with recurrent ovarian epithelial, peritoneal, or tubal cancer. II. Determine the nature and degree of toxicity of this treatment regimen in this patient population. III. Evaluate the response rate and time to disease progression in these patients.

OUTLINE: This is a dose escalation study. Patients receive oral topotecan daily on days 1-5 and oral etoposide daily on days 8-10. Courses repeat every 28 days in the absence of disease progression or unacceptable side effects. Patients achieving partial or complete response or stable disease continue treatment for at least 4-6 courses. Cohorts of 3-6 patients receive topotecan and etoposide on increasing numbers of days until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which no greater than 1 of 6 patients experiences dose limiting toxicity. Patients are followed every 3 months or until death.

PROJECTED ACCRUAL: A total of 24 patients will be accrued for this study within 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed ovarian epithelial, peritoneal, or tubal cancer Epithelial cell types Serous adenocarcinoma Endometrioid adenocarcinoma Mucinous adenocarcinoma Undifferentiated carcinoma Clear cell adenocarcinoma Mixed epithelial carcinoma Transitional cell Malignant Brenner's tumor Adenocarcinoma not otherwise specified Measurable or evaluable disease No brain or leptomeningeal metastases No symptomatic bowel involvement of ovarian cancer Not eligible for higher priority GOG phase II or III study

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: GOG 0-2 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 times normal SGOT/SGPT/GGT no greater than 3 times normal Alkaline phosphatase no greater than 3 times normal No acute hepatitis Renal: Creatinine no greater than 2.0 mg/dL OR Creatinine clearance greater than 50 mL/min Other: No septicemia or severe infection Body surface area at least 1 m2 Adequate intestinal function (i.e., does not require IV hydration or nutritional support) Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception 3 months prior to and during study No other malignancies within the past 5 years except curatively treated skin cancer No other severe medical problems that would prevent compliance No condition of the GI tract that would affect GI absorption and motility No severe gastrointestinal bleeding

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent immunotherapy Chemotherapy: No prior topotecan, other camptothecin analogs, or etoposide At least 1 prior cisplatin/paclitaxel based regimen At least 3 weeks since prior chemotherapy and recovered No more than 2 prior cytotoxic chemotherapy regimens No other concurrent chemotherapy Endocrine therapy: No concurrent hormonal therapy for cancer Radiotherapy: At least 3 weeks since prior radiotherapy to no more than 10% of the bone marrow and recovered No concurrent radiotherapy Surgery: Not specified Other: At least 28 days or 5 half lives since prior investigational drugs (including cytotoxic drugs) No concurrent metoclopramide or cisapride for maintaining gastric motility or emptying No chronic H2 antagonists, proton pump inhibitors, or antacids for gastritis, gastroesophageal reflux disease, or gastric or duodenal ulcers Intermittent antacids allowed, if no antacids 6 hours prior to and 90 minutes after topotecan

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 1999-09; Primary Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter G. Rose, MD, Study Chair — The Cleveland Clinic
Locations (6):
- United States (6):
  - Holden Comprehensive Cancer Center at The University of Iowa, Iowa City, Iowa
  - Mercy Medical Center, Inc., Baltimore, Maryland
  - Cooper Hospital/University Medical Center, Camden, New Jersey
  - Ireland Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio

REFERENCES:
- [Result] Rose PG, Markman M, Bell JG, Fusco NL. Sequential prolonged oral topotecan and prolonged oral etoposide as second-line therapy in ovarian or peritoneal carcinoma: a phase I Gynecologic Oncology Group study. Gynecol Oncol. 2006 Aug;102(2):236-9. doi: 10.1016/j.ygyno.2005.12.003. Epub 2006 Jan 18. PMID 16412499